CLINICAL TRIAL: NCT01042548
Title: Proteomics and Radiomics Research of Breast Cancer Markers in Tissue, Interstitial Fluid and Serum
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: David Scaife Foundation (Unknown)
Responsible Party: Principal Investigator, Min Sun, MD, PD, University of Pittsburgh
Other Study IDs: 09-028
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Proteomics; Breast Cancer Markers; Tissue Interstitial Fluid
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will be asked to allow us to collect an extra 2 tablespoons of blood at the time of pre-operative blood work. For those subjects with cancer who undergo surgery, a follow-up blood sample will be collected prior to chemotherapy, radiation, or hormonal therapy, and every six months afterwards at the time of their standard clinic/office visit for two years, then once a year for year 3-5. This will allow researchers to examine the samples to determine if blood changes over time after surgery, and what type of result may indicate a risk for recurrence.
  Any remaining blood samples not used for the study will remain in the laboratory for future research.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The current study is a case control study involving comparisons of tissue interstitial fluid from breast cancer and adjacent non-cancerous tissue as well as that from benign breast lesion and its adjacent non-diseased tissue for a distinguishable breast cancer profile. The purpose of this research is to collect fresh breast nodule/cancer and surrounding non-cancerous tissue for proteomic studies of the interstitial fluid to identify a profile distinguishing breast cancer which will also permit future research on stored interstitial fluid, blood or tissue samples. Specific markers identified from interstitial fluid study will be investigated in blood samples to develop serum markers for breast cancer diagnosis and prognosis. Additionally, we will perform both prospective and retrospective research on breast cancer involving clinical, demographic, epidemiologic information, treatment, follow-up and outcomes on breast nodule/cancer cases collected.

ELIGIBILITY:
Inclusion Criteria:

* All subjects ≥ 18 years of age undergoing surgery for indeterminate breast nodules, breast tissue reduction, prophylactic mastectomy, and all subjects with newly diagnosed invasive breast cancer will be eligible to participate. If invasive breast cancer or suspicion of invasive breast cancer, target lesion must measure ≥ 1.0 cm on breast imaging before core biopsy.

Exclusion Criteria:

* Anyone < 18 years of age.
* Multiple synchronous primary malignancies from different organ systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are receiving or seeking medical care at the UPMC St. Margaret for breast cancer will be invited to participate in the research study. Patients undergoing surgery for breast nodules suspected of being cancer or high risk lesions, breast tissue reduction, or prophylactic mastectomy will also be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-02-03 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC St. Margaret, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No